CLINICAL TRIAL: NCT03000543
Title: Validation of a Novel Isotope Dilution Technique to Assess Vitamin A Status in Infants
Brief Title: Novel Isotope Dilution Technique to Assess Vitamin A Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR-14126
Record Dates: First submitted 2016-12-14; First posted 2016-12-22 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2018-03

CONDITIONS: Healthy Infants; Infants With an Inflammatory Condition
Keywords: vitamin A; vitamin A isotope; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Vaccines; PENTA

ARMS (2):
- Vitamin A pool size in infants without inflammatory condition (No Intervention): Assessing vitamin A (VA) pool size in infants without inflammatory condition using model based compartmental analysis from the fraction of oral dose-derived 13C10-VA and 13C4-VA in plasma over time.
- Vitamin A pool size in infants with inflammatory condition (Experimental): Assessing vitamin A (VA) pool size in infants without inflammatory condition using model based compartmental analysis from the fraction of oral dose-derived 13C10-VA and 13C4-VA in plasma over time.
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Pentavalent vaccine. It is a combination of five different antigens (Hepatitis B (HBV)/ Haemophilus influenzae type b (HiB) / Tetanus-Diphtheria-whole cell Pertussis (TDwP)).
  Other Names: PENTA
  Arms: Vitamin A pool size in infants with inflammatory condition

SUMMARY:
Background:

There is no reliable method for vitamin A (VA) assessment for infants and young children. Serum VA concentration is not an authenticate indicator of VA status, while existing deuterium- VA isotope dilution methods to determine the whole body VA status require 3 weeks and not applicable for infants and children. The investigator's research group recently developed a new simplified equation to measure VA pool size in 4-5 days, correlated with compartmental model-predicted value and estimate VA pool size in adults with high precision. In this study, we validate the method in healthy infants and infants with an inflammatory condition.

Hypothesis:

Whole-body VA status in infant and children can be estimated without accounting for the fractional catabolic rate in the context of an inflammatory condition

Specific Objectives:

In this study, the investigators propose to determine the early time point equation for assessing VA pool size in infants with or without inflammatory condition using model-based compartmental analysis from the fraction of oral dose-derived 13C10-VA and 13C4-VA in plasma over time.

Methods:

A total of 183 infants (9-18 mo of age) will participate in this study in the following two phases of the "Super Kid study" that ensure no more than 2 venous blood samples from each infant, even though multiple time points (at least 4 subjects / time-point) over a 28-day study period will be available for mathematical modeling. In this study, investigators will use two different stable isotopic vitamin A e.g., 13C10-retinyl acetate and 13C4-retinyl acetate. 400 μg of these isotopes, dissolved in 0.5 mL of sunflower oil, will be provided directly into the infant's mouth by using a direct replacement pipette. Mothers will be asked to breastfeed their infant after oral dosing to enhance absorption of the labeled vitamin A. Specific activity of 13C10- and 13C4- retinyl acetate in the blood samples will be measured by liquid chromatography-tandem mass spectrometry (LC/MS/MS). Dietary and morbidity questionnaires will be used. Investigators will also use PENTA vaccines as a means to induce controlled inflammation (closely mimic to natural infection). PENTA is a combination of five different vaccine antigens (Hepatitis B (HBV)/ Haemophilus influenza type b (Hib) / Tetanus-Diphtheria-whole cell Pertussis (TDwP)). This vaccination is beneficial to the infants since the World Health Organization recommends a booster vaccination dose. At the end of the study, PENTA vaccines will also be provided to the study infants in the "no-vaccine" group.

(A) 115 infants will be enrolled randomly into 16 groups of them 40 infants will be in the first group, while other infants will be assigned in the other 15 groups (n=5/group). On day 0 (at 0h), all infants (n=115) will receive an oral dose of 13C10-retinyl acetate. Blood samples (5 mL) will be taken from 6h to 16th day of dosing at 9 different time-points. On day 16 (at 0h), randomly selected 50% infants (n=20) in the first group, as well as 30 infants in the other 6 groups, will receive PENTA vaccines, while the other 50% infants (n=20) in the first Group, as well as 45 infants in the other 9 groups, will receive no vaccines. 24 hours after vaccination (On day 17) a finger-prick blood sample will be obtained from the infants in the vaccinated group to measure CRP (QuikRead go, Orion, Finland). Infants who do not develop inflammation (CRP> 5mg/L) after PENTA vaccination will be excluded from the study. On day 17 (at 0h), all infants (n=115) will receive another oral dose of 13C4-retinyl acetate. Blood samples (5mL) will be collected from day 16 to day 28 at 11 different time-points for each of the vaccinated and non-vaccinated infants. This study will also assess the absorption of isotopic retinol by determining in total excreted stool up to 72 h post isotope dosing in a subsample of infants

(B) 68 infants will be enrolled in this phase. Of them, 28 infants will be assigned randomly into 7 groups (n=4/group). They will receive PENTA vaccines on day -1, and the next day (day 0) they will receive an oral dose of 13C4-retinyl acetate. Blood samples (5mL) will be collected from day 1 to day 28 at 8 different time points. In a separate design, 40 infants will receive an oral dose of 13C10-retinyl acetate on day 0 and blood samples (5mL) will be collected on day 4. On day 7 they all will receive another oral dose of 13C4-retinyl acetate (400 μg, dissolved in 0.5 mL of sunflower oil). On day 10, infants will receive PENTA vaccines (n=30) or no vaccine (n=10) and 1-day after vaccination, blood samples (5 mL) will be obtained from infants who develop inflammation (CRP> 5mg/L) in the vaccine group and also from infants in the control group (day 11).

Outcome measures:

The early time point equation for assessing VA pool size in a group of infants with or without inflammation

ELIGIBILITY:
Inclusion criteria:

1. 9 - 18 months of age
2. Infants with normal body temperature and normal CRP (<5 mg/L)
3. Infants receive breast milk from the mother at least once per day
4. Mothers produce a breast milk containing 30-40 nmol vitamin A /g milk fat
5. Infants received a high-dose vitamin A capsules at the time of the most recent national distribution campaign (within the last 2-4 months)
6. Mother is 18 - 45 years of age
7. Mother and her infant plan to stay in the study area for the duration of the study

Exclusion criteria:

1. Mother or infant has chronic disease
2. Mother or infant has acute illness on the day of data collection
3. Infant is anemic (Hb <90 g/L)
4. Infant has weight for length <80% of the reference median
5. Infants do not develop inflammation (CRP ≥5 mg/L) after PENTA vaccination

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Vitamin A pool size in infants with or without inflammation | Kinetic study for 28 days for each of the 2 groups of infants

CONTACTS AND LOCATIONS:
Overall Officials: Shaikh M Ahmad, Ph.D., Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (2):
- Bangladesh (2):
  - Clinical Trail Unit (CTU), icddr,b., Dhaka
  - Shaikh Meshbahuddin Ahmad, Dhaka

REFERENCES:
- [Derived] Ford JL, Green JB, Haskell MJ, Ahmad SM, Mazariegos Cordero DI, Oxley A, Engle-Stone R, Lietz G, Green MH. Use of Model-Based Compartmental Analysis and a Super-Child Design to Study Whole-Body Retinol Kinetics and Vitamin A Total Body Stores in Children from 3 Lower-Income Countries. J Nutr. 2020 Feb 1;150(2):411-418. doi: 10.1093/jn/nxz225. PMID 31535129